CLINICAL TRIAL: NCT00752362
Title: PercutAneous INTervention With Biodegradable- Polymer Based Paclitaxel-eluting, Sirolimus-eluting, or Bare Stents for the Treatment of de Novo Coronary Lesions.
Brief Title: Per-cutaneous Intervention Based Paclitaxel and Sirolimus-Eluting Versus Bare Stents for the Treatment of de Novo Coronary Lesions (PAINT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: CMS Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The PAINT Trial
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Restenosis
Keywords: Supralimus®,; Infinnium®,; Matrix®,; Restenosis; Percutaneous; Revascularization; Techniques; Metallic; Platform; Agents; Antiproliferative; Properties
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Percutaneous coronary intervention with bare metal stent
  Interventions: Device: Milennium Matrix® (Control)
- 2 (Experimental): Percutaneous coronary intervention with paclitaxel-eluting stent
  Interventions: Device: Infinnium®
- 3 (Experimental): Percutaneous coronary intervention with sirolimus-eluting stent
  Interventions: Device: Supralimus®

INTERVENTIONS:
Device: Milennium Matrix® (Control) — Percutaneous coronary intervention with bare metal stent
  Other Names: Milennium Matrix®
  Arms: 1
Device: Infinnium® — Percutaneous coronary intervention with paclitaxel-eluting stent
  Arms: 2
Device: Supralimus® — Percutaneous coronary intervention with sirolimus-eluting stent
  Arms: 3

SUMMARY:
Objectives:

PRIMARY OBJECTIVE:

To compare the in-stent late loss at 9 months of paclitaxel- and sirolimus- eluting stents with the late loss of bare metal control stents.

SECONDARY OBJECTIVES:

Safety:

To compare the occurrence of Major Adverse Cardiac Events (MACE) at 30 days, 9 months, 1 year, 3 years and 5 years among the paclitaxel, sirolimus and control study arms.

To compare the occurrence de Serious Adverse Events (SAEs) within 5 years among the paclitaxel, sirolimus and control study arms.

To compare the occurrence of in-stent thrombosis within 5 years among the paclitaxel, sirolimus and control study arms.

Efficacy:

To compare the rate of angiographic success among the study groups To compare the rate of procedural success among the study groups To compare the incidence of clinically driven target lesion revascularization at 9 months, 1 year, 3 years and 5 years among the paclitaxel, sirolimus and control study arms.

To compare the incidence of clinically driven target vessel revascularization at 9 months, 1 year, 3 years and 5 years among the paclitaxel, sirolimus and control study arms.

To compare the 1-year, 3-year and 5-year cost-effectiveness profile of the paclitaxel, sirolimus and control study arms.

To compare the 9-month in-stent late loss of paclitaxel-eluting stents to the in-stent late loss of sirolimus-eluting stents To compare the 9-month in-segment late loss among the study groups To compare the 9-month in-stent and in-segment binary restenosis rate among the study groups To compare the IVUS percent neointimal obstruction among the study groups

Study Design:

In the present RANDOMIZED study, the paclitaxel-eluting stent Infinnium® and the sirolimus-eluting stent Supralimus® will be compared to a metallic stent with the same structure (Milennium Matrix®) but without drug elution for the treatment of de novo lesions in native coronaries. The study will be a multicenter clinical trial and will include patients for the treatment with one of the three study stents. In total, 275 patients will be enrolled, randomly allocated for the Infinnium®, Supralimus®, or Milennium Matrix® stents in a 2:2:1 proportion. Patients will be followed-up for 12 months after the index procedure. All patients will undergo a follow-up angiography at 9 months. A subgroup of 55 patients will be evaluated at 9 months with IVUS examination.

Treatment:

Patients will be treated, according to the randomization groups, with Infinnium®, Supralimus®, or Milennium Matrix® stents of 19 mm, 23 mm, or 29 mm and nominal diameters of 2.5, 3.0, and 3.5 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Symptomatic ischemic heart disease and/or objective evidence of myocardial ischemia;
3. De novo coronary lesion (non-restenosis);
4. Target lesion located in a native artery;
5. Target lesion located in a vessel with diameter between 2.5-3.5 mm (visual analysis);
6. Target lesion amenable to treatment with a single stent of up to 29 mm in length;
7. Target lesion with a diameter stenosis > 50% (visual analysis);
8. Acceptable candidate for surgical revascularization;
9. Signed informed consent term.

Exclusion Criteria:

GENERAL EXCLUSION CRITERIA

1. Q-wave myocardial infarction < 48 hours before the index procedure
2. Recent myocardial infarction, with or without Q waves, with cardiac markers levels still above the normal upper limits
3. Left ventricle ejection fraction ≤30%
4. Renal dysfunction (serum creatinine > 2.0 mg/dl [>177 µmol/l])
5. Platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3
6. White cell count < 3.000 cells/mm3
7. Suspected or known liver disease (including subclinical hepatitis)
8. Heart transplant recipient
9. Know allergy to aspirin, clopidogrel, ticlopidine, paclitaxel, sirolimus, heparin, or stainless steel
10. Life expectancy < 12 months
11. Any medical condition that, in the opinion of the investigator, may interfere with the ideal participation in study
12. Current inclusion in another study to investigate drug or other device, or planned inclusion in another study to investigate drug or other device during the follow-up.
13. Coronary angioplasty (with or without stent) < 6 months in any segment of the target vessel
14. Previous coronary angioplasty (with or without stent), at any time, in a coronary segment < 5 mm (proximal or distal) from the target lesion
15. Coronary angioplasty (with or without stent) in any segment of the target vessel planned during the next 12 months following the index procedure.

ANGIOGRAPHIC EXCLUSION CRITERIA

1. Restenotic target lesion
2. Need for treatment of more than one lesion in the target vessel;
3. Diameter of the target vessel < 2.5 mm or > 3.5 mm (visual analysis)
4. Long target lesion, not amenable to treatment with a single stent of up to 29 mm in length, according to the operator's discretion
5. Significant (> 50%) unprotected left main lesion
6. Angiographic thrombus
7. Target lesion located in bypass graft
8. Occluded target vessel (antegrade flow TIMI 0 or 1)
9. Target lesion in ostial location;
10. Target lesion in a bifurcation site with a side branch > 2.5 mm or that may require stent implantation;
11. Calcified target lesion with anticipated unsuccessful balloon pre-dilatation;
12. Severely tortuous target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
compare the in-stent late loss at 9M of paclitaxel- and sirolimus- eluting stents with the late loss of bare metal control stents. | 9 months

SECONDARY OUTCOMES:
MACE at 1,9&12M, SAE & ST until 12M. Rate of angiographic & procedural success, TLR & TVR at 1&9M Instent LL between Supralimus®, Infinnium® & Matrix® Insegment binary restenosis at 9M IVUS% neointimal obstruction cost-effectiveness profile at 12M | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Pedro A. Lemos, MD, Principal Investigator — Instituto do Coração - InCor
Locations (11):
- Brazil (11):
  - Hospital Universitário Walter Cantídio, Fortaleza, Ceará
  - Hospital Universitário Cassiano Antonio de Moraes, Vitória, Espírito Santo
  - Hospital Meridional Intercath, Vitória, Espírito Santo
  - Hospital Biocor, Belo Horizonte, Minas Gerais
  - Rede D'Or de Hospitais, Rio de Janeiro, Rio de Janeiro
  - Hospital Natal Center, Natal, Rio Grande do Norte
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital São Paulo - UNIFESP, São Paulo, São Paulo
  - Hospital São Camilo, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Instituto do Coração - InCor, São Paulo

REFERENCES:
- [Result] Lemos PA, Moulin B, Perin MA, Oliveira LA, Arruda JA, Lima VC, Lima AA, Caramori PR, Medeiros CR, Barbosa MR, Brito FS Jr, Ribeiro EE, Martinez EE; PAINT study. Rationale and design for the PAINT randomized trial. Arq Bras Cardiol. 2009 Dec;93(6):547-53, 590-7. doi: 10.1590/s0066-782x2009001200006. English, Portuguese. PMID 20379631
- [Result] Lemos PA, Moulin B, Perin MA, Oliveira LA, Arruda JA, Lima VC, Lima AA, Caramori PR, Medeiros CR, Barbosa MR, Brito FS Jr, Ribeiro EE, Martinez EE; PAINT trial investigators. Randomized evaluation of two drug-eluting stents with identical metallic platform and biodegradable polymer but different agents (paclitaxel or sirolimus) compared against bare stents: 1-year results of the PAINT trial. Catheter Cardiovasc Interv. 2009 Nov 1;74(5):665-73. doi: 10.1002/ccd.22166. PMID 19670303
- [Result] Lemos PA, Moulin B, Perin MA, Oliveira LA, Arruda JA, Lima VC, Lima AA, Caramori PR, Medeiros CR, Barbosa MR, Brito FS Jr, Ribeiro EE. Late clinical outcomes after implantation of drug-eluting stents coated with biodegradable polymers: 3-year follow-up of the PAINT randomised trial. EuroIntervention. 2012 May 15;8(1):117-9. doi: 10.4244/EIJV8I1A18. PMID 22580255
- [Result] Marchini JF, Gomes WF, Moulin B, Perin MA, Oliveira LA, Arruda JA, Lima VC, Lima AA, Caramori PR, Medeiros CR, Barbosa MR, Brito FS Jr, Ribeiro EE, Lemos PA. Very late outcomes of drug-eluting stents coated with biodegradable polymers: insights from the 5-year follow-up of the randomized PAINT trial. Cardiovasc Diagn Ther. 2014 Dec;4(6):480-6. doi: 10.3978/j.issn.2223-3652.2014.12.05. PMID 25610805